CLINICAL TRIAL: NCT05044091
Title: Homologous Recombination Deficiency Associated With Response to Poly (ADP-ribose) Polymerase Inhibitors in Ovarian Cancer Patients: the First Real-word Evidence From China
Brief Title: Homologous Recombination Deficiency in Chinese Ovarian Cancer Patients
Acronym: HOPEI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiaoxiang Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaoxiang Chen, Academic secretary of gynecological oncology Committee of Jiangsu anti cancer association, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Other Study IDs: JiangsuCIH010
Record Dates: First submitted 2021-09-04; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Cancer; HRD; PARP Inhibitor
Keywords: Ovarian caner, HRD, PARP inhibitor
MeSH Terms: conditions — Ovarian Neoplasms; Kenny-Caffey syndrome, Type 1 | interventions — Poly(ADP-ribose) Polymerase Inhibitors; olaparib; niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The formalin fixation and paraffin embedding (FFPE ) samples from the cytoreductive surgery will be obtained after patients' informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ovarian/fallopian tube/primary peritoneal cancer patients: ovarian/fallopian tube/primary peritoneal cancer patients treated with PAPRi for more than four weeks
  Interventions: Drug: PARP inhibitor

INTERVENTIONS:
Drug: PARP inhibitor — Ovarian/fallopian tube/primary peritoneal cancer patients with PARP inhibitors according to the NCCN guideline and their instructions
  Other Names: Lynparza, Zejula

SUMMARY:
Homologous recombination deficiency (HRD) is an important molecular biomarker for Poly (ADP-ribose) polymerase inhibitors (PARPi) which is a significant progress in the treatment of ovarian cancer. However, the proportion of HRD positive in real world and relationship of HRD status with PARPi in Chinese ovarian cancer patients remains unknown.

DETAILED DESCRIPTION:
This study intends to perform HRD testing of ovarian cancer in real world from China and correlate HRD status and clinical characteristics with therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects join the study voluntarily and sign informed consent;
2. Female subjects are older than 18 years;
3. ECOG(Eastern Cooperative Oncology Group) physical status score is 0-2;
4. Life expectancy≥3 months;
5. Histologically confirmed FIGO(International Federation of Gynecology and Obstetrics ) III/IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer; Participants must have high-grade serous or endometrioid histology;
6. Patients received PARP inhibitor as maintenance therapy or monotherapy for more than four weeks.

Exclusion Criteria:

1. Personnel involved in the formulation or implementation of the research plan;
2. Patient participated in other clinical trails using other experimental drugs at the same time as the study;
3. The subjects had other malignant diseases in past 2 years, except skin squamous cell carcinoma, basal-like carcinoma, breast intraductal carcinoma in situ, or cervical carcinoma in situ;
4. Previous or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
5. Patients who are pregnant or lactation, or who plan to become pregnant during study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian/fallopian tube/primary peritoneal cancer patients treated with PARP inhibitor in the real word.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average of 1 year
  ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR) as assessed by RECIST1.1.
Progression Free Survival (PFS) | Through study completion, an average of 1 year
  PFS is defined as the time in months from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death as assessed by RECIST1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiang Chen, MD,PhD, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (1):
- Xiaoxiang Chen, MD,PhD, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Chen and Dr. Ni for primary data.